CLINICAL TRIAL: NCT00803582
Title: Effectiveness of Acupuncture for Phonotraumatic Injuries
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Prof Edwin Yiu, The University of Hong Kong
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT003879 (NIH); R21AT003879 (NIH); Acu_R21_1
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2010-01

CONDITIONS: Phonotraumatic Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Experimental (Experimental): Traditional acupuncture
  Interventions: Procedure: Traditional Chinese acupuncture
- Placebo (Sham Comparator): Placebo acupuncture
  Interventions: Procedure: Placebo acupuncture
- No-treatment (No Intervention): no treatment

INTERVENTIONS:
Procedure: Traditional Chinese acupuncture — Acupuncture at two Hegu (LI4) and two Lieque (Lu7) points on the wrist, one Lianquan (CV23) and two Renying (St9) points on the neck and two Zhaohai (Ki6) for 12 30-minute sessions
  Other Names: Ordinary acupuncture
  Arms: Experimental
Procedure: Placebo acupuncture — Placebo acupuncture at two Hegu (LI4) and two Lieque (Lu7) points on the wrist, one Lianquan (CV23) and two Renying (St9) points on the neck and two Zhaohai (Ki6) for 12 30-minute sessions.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy of acupuncture for the treatment of phonotraumatic lesions of the vocal folds, using the International Classification of Functioning Disability and Health (World Health Organization, 2001) as the conceptual framework to guide the selection of outcome measures.

DETAILED DESCRIPTION:
The experimental hypothesis for this study is that needling at the designated treatment acupoints will bring about greater improvement in structural and functional impairment in the vocal folds and its sequelae, as compared to placebo treatment. However, it is further hypothesized that treatment benefits from acupuncture will be outweighed by continued phonotrauma following termination of treatment, and thus will not be maintained at long-term follow-up. Further, it is expected that voice-related quality-of-life improvements may be equal for genuine acupuncture as compared to placebo. Finally, it is hypothesized that the acupuncture protocol should have comparable effects for male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Otolaryngological diagnosis within the preceding 15 days of swelling or thickening of at least one vocal fold, or nodules, fibrous mass, cyst, polyp, or chronic (non-infectious) laryngitis, which by history are traceable to phonotrauma and by history appear stable or worsening;
2. age 20-55 yr

Exclusion Criteria:

1. no prior voice therapy;
2. no medication or therapy that may affect voice during the period of participation;
3. no acupuncture treatment for any condition within the preceding 10 year;
4. no diagnosed or suspected neurological conditions, hearing loss (i.e. hearing threshold of the better ear not exceeding 35dB HL at 250 Hz, 500 Hz, 1000 Hz, 4000 Hz and 8000 Hz), history of asthma, and no upper respiratory infection at the time of recruitment.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Estimated)
Dates: Start 2007-02; Primary Completion 2010-02 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Maximum fundamental frequency of the voice range profile | Pre-treatment, Mid-treatment, Post-treatment, 2 weeks post-treatment, 4 weeks post-treatment, 3 months post-treatment

SECONDARY OUTCOMES:
Voice Activity and Participation Profile | Pre-treatment, Mid-treatment, Post-treatment, 2 weeks post-treatment, 4 weeks post-treatment, 3 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Yiu, Prof, Principal Investigator — The University of Hong Kong
Locations (1):
- Voice Research Laboratory, The University of Hong Kong, Hong Kong, Hong Kong